CLINICAL TRIAL: NCT02260414
Title: Effects of Injection Tinzaparin Prophylactic Dose (4,500 IU Anti-Xa) on Thrombin Generation in Patients With Multiple Myeloma, Lymphoma Patients and Patients Hospitalized for an Acute Medical Condition.
Brief Title: Effects of Anticoagulant Preventive Injection in Patients With Blood Cancer
Acronym: METRO B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1408049; 2014-000946-31 (EudraCT Number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-09 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma; Multiple Myeloma
Keywords: Endogenous Thrombin Potential; Lymphoma; Multiple Myeloma; tinzaparin; thrombin generation; Thromboplastin generation tests
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Tinzaparin; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with multiple myeloma (Experimental): Patient with multiple myeloma indication with de novo standard treatment thalidomide or lenalidomide or erythropoietin treated with one injection of 4500 IU tinzaparin and blood samples taken at hours : 0, 3, 8, 18 and 24 after subcutaneous injection of tinzaparin
  Interventions: Drug: Tinzaparin; Other: Blood sample
- Patients with agressive lymphoma (Active Comparator): Patient hospitalized for aggressive lymphoma treated with chemotherapy treated with one injection of 4500 IU tinzaparin and blood samples taken at hours : 0, 3, 8, 18 and 24 after subcutaneous injection of tinzaparin
  Interventions: Drug: Tinzaparin; Other: Blood sample
- Patients with acute medical condition (Active Comparator): Patient older than 40 years and hospitalized at least three days for an acute medical pathology type of acute respiratory or cardiac treated with one injection of 4500 IU tinzaparin and blood samples taken at hours : 0, 3, 8, 18 and 24 after subcutaneous injection of tinzaparin
  Interventions: Drug: Tinzaparin; Other: Blood sample

INTERVENTIONS:
Drug: Tinzaparin — single subcutaneous injection of 4500 IU tinzaparin
Other: Blood sample — blood sample taken at hours 0, 3, 8, 18 and 24 after subcutaneous injection of 4500 IU tinzaparin

SUMMARY:
In cancer, the incidence of venous thromboembolism (VTE) is particularly high in patients with myeloma, especially when it is de novo and treated with thalidomide, lenalidomide or erythropoietin. Curiously, the prevention of VTE with LMWH (low-molecular-weight heparin) in myeloma seems no more effective than that achieved with aspirin, while the effectiveness of the latter in the primary prevention of VTE has never been demonstrated regardless of the type of population considered. Meanwhile, a biological study showed that prophylactic doses of LMWH in patients with different types of cancer did not always optimal reduction of thrombin peak during the 24 hours following the injection of LMWH. These clinical and biological studies lead to the conclusion that patients with myeloma may be resistant to the usual doses of preventive LMWH, which may explain the failure of prevention.

Initially we intend to investigate whether this resistance to prophylactic doses of LMWH is present in patient's biology and if this resistance is specific to myeloma in hematological cancers. For this, we propose to study the evolution of thrombin generation by Thrombinography during 24 hours after subcutaneous injection of 4500 anti-Xa IU Tinzaparin in 6 patients with de novo myeloma whit high thrombo embolic risk ie treated with thalidomide, lenalidomide or erythropoietin. LMWH is Tinzaparin chosen because it does not accumulate in patients with impaired renal function, and has a greater anti-biological activity thrombotic than other LMWH.

To assess whether the observed pattern of thrombin generation is particularly multiple myeloma, we will take the same study in 6 patients with aggressive lymphoma and 6 medical patients hospitalized for acute heart and respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight between 40 and 100 kg
2. Patient:

2a- With multiple myeloma indication with de novo standard treatment thalidomide or lenalidomide or erythropoietin (group 1) 2b- Or hospitalized for aggressive lymphoma treated with chemotherapy (group 2) 2c- Or older than 40 years and hospitalized at least three days for an acute medical pathology type of acute respiratory or cardiac (group 3) decompensation

Exclusion Criteria:

* Patient requiring anticoagulant therapy at curative doses
* Patients with a lower platelet count 80 G / L
* Subject with a history of heparin-induced thrombocytopenia
* Subject with a history of hemorrhagic disease
* History of severe trauma within 6 weeks prior to enrollment
* Organic lesion at risk of bleeding
* Poor renal with creatinine clearance <30 ml / min
* Hypersensitivity to Tinzaparin
* Events or bleeding tendencies associated with coagulation disorders
* Subject on oral anticoagulant
* For group 3: Presence of hematological malignancy or active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Endogenous Thrombin Potential (ETP, nM.min) for all patients with de novo myeloma with high thrombotic risk | hours : 0, 3, 8, 18, 24
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Tests (TGTs) following a single injection of 4500 IU tinzaparin

SECONDARY OUTCOMES:
Endogenous Thrombin Potential (ETP, nM.min) for all patients with aggressive lymphoma treated with chemotherapy | hours : 0, 3, 8, 18, 24
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Tests (TGTs) following a single injection of 4500 IU tinzaparin
Endogenous Thrombin Potential (ETP, nM.min) for all patients with over 40 years hospitalized for heart or respiratory failure | hours : 0, 3, 8, 18, 24
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Tests (TGTs) following a single injection of 4500 IU tinzaparin
Differences of Endogenous Thrombin Potential (ETP, nM.min) between group 1 and group 2 et 3 | hours : 0, 3, 8, 18, 24
  Endogenous Thrombin Potential (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Tests (TGTs) following a single injection of 4500 IU tinzaparin

CONTACTS AND LOCATIONS:
Overall Officials: Bernard TARDY, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France